CLINICAL TRIAL: NCT02979860
Title: Experimental Changes in Children's Sleep Duration and Timing: Effect on Obesity and Type 2 Diabetes Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 24131
Record Dates: First submitted 2016-11-29; First posted 2016-12-02 (Estimated); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Type2 Diabetes; Sleep
MeSH Terms: interventions — Sleep Duration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Typical sleep schedule (No Intervention): Children in this arm will be asked to maintain their current sleep schedule. No prescription will be provided other than to sleep how they "typically" would sleep.
- Enhance time in bed by 90 min/night (Experimental): Sleep duration - 90 minutes: Children in this arm will be asked to get into bed and to turn their lights out 90 minutes earlier than their typical bedtime. Bedtimes and wake times will remain consistent across the 4-week experimental phase of the study.
  Interventions: Behavioral: Sleep duration 90 min
- Enhance time in bed by 45 min/night (Experimental): Sleep duration - 45 minutes:Children in this arm will be asked to get into bed and to turn their lights out 45 minutes earlier than their typical bedtime. Bedtimes and wake times will remain consistent across the 4-week experimental phase of the study.
  Interventions: Behavioral: Sleep duration 45 min
- Regularize sleep schedule (Experimental): Sleep timing: Children in this arm will be asked to get into bed at a consistent bedtime each night and wake at a consistent time each morning such that time in bed achieved during baseline is maintained during the 4-week experimental phase; only timing of bedtimes/wake times will be manipulated in this arm.
  Interventions: Behavioral: Sleep timing

INTERVENTIONS:
Behavioral: Sleep duration 90 min — Sleep duration: time in bed increased by 90 minutes
  Arms: Enhance time in bed by 90 min/night
Behavioral: Sleep duration 45 min — Sleep duration: time in bed increased by 45 minutes
  Arms: Enhance time in bed by 45 min/night
Behavioral: Sleep timing — Sleep timing: bed time kept consistent
  Arms: Regularize sleep schedule

SUMMARY:
Enhancing children's sleep duration and/or timing may represent a novel approach for weight regulation and prevention of T2DM. The proposed study will assess how experimental changes in children's sleep duration and timing affect weight regulation and T2DM risk. Sixty African American children ages 8-11 years old who sleep approximately 9.5 hours or less each night will be enrolled into a 4-arm randomized controlled pilot to compare three experimental manipulations in children's sleep to a "typical sleep" (TYP) control. Experimental arms will include: 1) increase in time in bed (TIB) by 90 minutes/night; 2) increase in TIB by 45 minutes/night; or 3) consistent (CON) sleep schedule (but no change in TIB). At baseline, 2- and 4-week follow-up, participants be weighed and measured for height, have body fat assessed (bod pod), and their blood drawn (following an overnight fast). The pilot will provide important data on the potential role of sleep in combating disparities in cardiometabolic risk. Primary aims are: 1) to determine the effects of changes in sleep on changes in glucose regulation and 2) to determine the effect of changes in sleep on additional measures of glucose regulation and adiposity.

DETAILED DESCRIPTION:
Eligible families who provide consent/assent will be enrolled into a five week study. All families will complete assessments at baseline, two weeks and four weeks. Each assessment lasts one week and children will be asked to wear an actigraph on their wrist (to measure sleep) and an accelerometer on their hip (to measure physical activity). At the end of the week families will be scheduled for a visit at the research center first thing in the morning approximately one hour after waking and following an overnight fast. During this visit, actigraphs and accelerometers will be downloaded and data will be reviewed with families. Children will be weighed and measured for height and have their body composition assessed. To measure glucose regulation, children will first have 5 ml of blood drawn in a fasted state. They will then ingest a glucose solution (1.75 g/kg; maximum of 75 g) over 2 minutes, and blood will be drawn (1.5 ml) 120 min after the child consumes the solution. At week 4, 5 ml blood will be drawn fasting; OGTT will not be administered (see note below). Research staff will also complete one-day dietary recalls with participants at each center-based assessment to obtain information on all foods consumed over the previous 24-hour period. In addition, at the baseline assessment only, parents will complete questionnaires on basic demographic information and child sleep. It is anticipated that the total time for each assessment will take approximately 2.5-3 hours (1 hour at 4 weeks). Following eligibility confirmation at the baseline assessment, families will be randomized to one of four protocols: 1) Enhance TIB by 90 min/night; 2) Enhance TIB by 45 min/night; 3) Regularize Sleep Schedule; or 4) Typical Sleep Schedule.

Continuous glucose monitoring In a voluntary subset of randomly selected children (approximately n = 4/group) 72-hour continuous glucose monitoring (CGM) will be performed. If the child and family agree to participate in CGM, they will come to the Center for an additional visit during which a disposable subcutaneous glucose-sensing device connected to a battery-operated recorder will be inserted subcutaneously (a thin tube under the surface of the skin). This sensor measures glucose every ten seconds and records an average value every five minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Parent-reported child race African American/Black.
2. Parent-reported child age of 8-11 years
3. Less than or equal to approximately 9.5 hours time in bed (TIB; based on actigraphy and sleep diaries)
4. Variability in Sleep Patterns (based on actigraphy and sleep diaries)
5. BMI for age and gender > 85th percentile (but no greater than 100% overweight)
6. Self-reported parent age of 18 years, primary caretaker, and at home throughout the study (i.e., at bedtimes and wake times)
7. Reported willingness to complete all study tasks, including blood draws

Exclusion Criteria:

1. Diagnosable Sleep Disorder
2. Parent-reported diagnosis of medical or psychiatric condition that may impact sleep/weight status
3. Actively trying to lose weight
4. Inability to Understand or Complete Protocol
5. Sibling of enrolled subjects

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2021-04-08 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Insulin Resistance | 4 weeks
  Fasting plasma insulin and glucose will be used to compute the homeostatic model assessment of insulin resistance (HOMA-IR).

SECONDARY OUTCOMES:
Metabolic Measures | 3 3-hour assessment visits
  Blood will be drawn before and after the consumption of a glucose solution to compute an Insulin Sensitivity Index (ISI) and glucose tolerance.

OTHER OUTCOMES:
Anthropometrics | 3 3-hour assessment visits
  Child weight will be obtained on a digital scale and height on a wall-mounted stadiometer using standard procedures and while in street clothes, without shoes. Measures will be converted to BMI, BMIz, and BMI percentile using age and sex-adjusted normative data from the CDC.
Body Composition | 3 3-hour assessment visits
  Youth body composition (% body fat) will be estimated by air displacement plethysmography (BOD POD®; Life Measurement Instruments, Concord, CA).
Acceptability/Feasibility | 2 3-hour assesment Visit
  Acceptability and feasibility of each experimental approach for changing sleep will be assessed with semi-structured qualitative interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Chantelle Hart, PhD, Principal Investigator — Temple University
Locations (1):
- Center for Obesity Research and Education, Temple University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No